CLINICAL TRIAL: NCT05257928
Title: Evaluation of a Carepartner-Integrated Telehealth Gait Rehabilitation Program for Persons With Stroke
Brief Title: Carepartner Collaborative Integrated Therapy Gait (CARE-CITE-Gait) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Principal Investigator, Sarah Blanton, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004000
Record Dates: First submitted 2022-02-11; First posted 2022-02-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Telehealth; Rehabilitation; Care partner; Sub-acute stroke; CARE-CITE Gait; Stroke survivors; Caregiver
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE-CITE GAIT Carepartner (Experimental): This study arm consists of carepartners (CP) receiving the CARE-CITE Gait intervention. Over a period of one month, alongside the stroke survivor, the CP will receive 2 two-hour home-based therapy visits with a licensed physical therapist to develop therapy goals related to gait, mobility and balance and develop a home exercise plan to improve function. The CP will receive two additional phone calls to discuss the online CARE-CITE educational modules.
  Interventions: Behavioral: CARE-CITE Gait
- CARE-CITE GAIT Stroke Survivor (Experimental): This study arm consists of stroke survivors (SS) of carepartners receiving the CARE-CITE Gait intervention. Over a period of one month, along with the CP, the SS will receive 2 two-hour home-based therapy visits with a licensed physical therapist to develop therapy goals related to gait, mobility and balance and develop a home exercise plan to improve function.
  Interventions: Behavioral: CARE-CITE Gait

INTERVENTIONS:
Behavioral: CARE-CITE Gait — The CARE-CITE intervention content modified to address gait rehabilitation, and test 4-weeks of CARE-CITE-Gait in 15 CP/SS dyads.It will occur in the dyad's home.CP will complete 6 online CARE-CITE modules. Modules will include demonstration videos and instructive content covering the following areas:principles of functional task practice, the adaptation of tasks, and importance of progression of challenging tasks to drive neuroplasticity. Examples are provided to address potential SS frustration and improve adherence.Underpinning the content is the concept of autonomy support,with examples of fostering empathy, problem-solving, instruction in the use of non-controlling language with role-playing situations and the importance of creating choice in activities. During the two home therapy sessions, the physical therapist will work with the CP and stroke survivor to collaboratively develop goals and an exercise program to improve mobility, gait and balance.

SUMMARY:
Stroke affects both the carepartner (CP) and stroke survivor (SS), with CPs frequently feeling overwhelmed and exhausted. The investigators have developed a theory-based, family-centered intervention, Carepartner Collaborative Integrated Therapy (CARE-CITE) designed to positively engage CPs during SS daily activities and rehabilitation exercise practice in the home setting. Using a web-based program with exemplary interactive videos of family scenarios in the home, CARE-CITE guides the CP in collaborative goal setting and creating an autonomy-supportive environment with the SS to promote motivation and creative problem-solving.

This study will use the modified upper extremity-focused CARE-CITE intervention content to address gait rehabilitation, and test 4-weeks of CARE-CITE-Gait in 15 CP/SS dyads to determine if similar positive outcomes are seen with integration to gait rehabilitation. Over a period of one month, SS and CP will receive 2 two-hour home-based therapy visits with a licensed physical therapist to develop therapy goals related to gait, mobility and balance and develop a home exercise plan to improve function. The CP will receive two additional phone calls to discuss the online CARE-CITE educational modules. The overall impact of this work is the development of innovative family-centered telerehabilitation interventions to improve self-management and physical activity.

DETAILED DESCRIPTION:
Stroke affects both the carepartner (CP) and stroke survivor (SS), with CPs frequently feeling overwhelmed and exhausted. Rehabilitation therapy activities largely do not address CP's well-being. The investigators have developed a theory-based, family-centered intervention, Carepartner Collaborative Integrated Therapy (CARE-CITE) designed to positively engage CPs during SS daily activities and rehabilitation exercise practice in the home setting. Using a web-based program with exemplary interactive videos of family scenarios in the home, CARE-CITE guides the CP in collaborative goal setting and creating an autonomy-supportive environment with the SS to promote motivation and creative problem-solving. To date, CARE-CITE has been evaluated in SS with chronic stroke and coupled with upper extremity therapy interventions. Promising preliminary data showed improvement in CP psychosocial outcomes and SS upper extremity function. The potential impact of CARE-CITE on SS mobility and gait recovery is unknown.

The investigators now seek to broaden the scope of the intervention by pairing CARE-CITE with home-based gait and functional mobility training (CARE-CITE-Gait). The goal of this proposal is to assess the impact of a novel home-based CARE-CITE-Gait intervention using a user-friendly telehealth delivery system. Aim 1 will evaluate usability, acceptability, and feasibility of CARE-CITE-Gait. Aim 2 will use a single site, quasi-experimental design with repeated measures (two baseline visits, post, and 1-month follow-up) to test 4-weeks of CARE-CITE-Gait in 15 CP/SS dyads to determine if similar positive outcomes are seen. Wearable sensors will be used to evaluate physical activity within the home and community. These data will support a larger randomized controlled trial testing the CARE-CITE-Gait intervention.

Study participants will be identified and recruited with successful techniques established by the PI (Blanton) and Co-I (Kesar) within the Emory Healthcare system and regional Atlanta hospitals, partnering with clinical staff for referrals and meeting with local stroke support groups. All Emory Rehabilitation Hospital stroke admissions will be screened based upon study inclusion/exclusion criteria and contacted by the research coordinator, if eligible. Participant eligibility will be confirmed via telephone screen, and initial clinical evaluation will follow at the Emory Rehabilitation Clinic. Eligible dyads (CP and SS) will be consented and evaluated at Emory Rehabilitation Hospital. Administration of CARE-CITE Gait intervention will occur in participants' homes over a period of 4 weeks, which includes CP review of the online CARE-CITE Gait education modules, two 2-hour home visits and 2 telerehabilitation check in video conference calls. All dyads will receive compensation for study participation at the end of the 1-month follow-up or prorated based on completed study evaluations.

The overall impact of this work is the development of innovative family-centered telerehabilitation interventions to improve self-management and physical activity. By providing a family-focused approach to gait and physical activity interventions, this project will help develop more effective treatments that improve both carepartner and stroke survivor outcomes after stroke.

ELIGIBILITY:
Inclusion Criteria:

* All SSs will be >3 months post-ischemic or hemorrhagic event, discharged from inpatient neurologic rehabilitation to their home, able to walk 10-meters with or without an assistive device, no severe cognitive deficits, no physician determined major medical or musculoskeletal problems that would limit participation, and a CP living in the home.
* CPs must be >21 years old, able to read and write English and have no significant cognitive deficits. CPs will be defined as those individuals who are a spouse/partner or family member dwelling in the same household. CPs must be familiar with using a computer and accessing websites or be familiar with using a tablet (available for loan if no computer is available).

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Individuals who are not able to clearly understand English
* Community Participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 month post intervention
  Recruitment rates will be calculated based on the percentage of those participants enrolled and randomized from those screened. Recruitment will be deemed feasible if the target enrollment of 15 dyads (2-3 dyads per month) is reached during the study timeframe.
Retention rate | 1 month post intervention
  Retention of participants will be tracked, recording the percentage of dropouts. Lower percentage correlates with better outcome.
Carepartners adherence rate | 1 month post intervention
  Carepartners (CP) adherence will be measured by the number of modules reviewed (6 total modules). Higher number indicates better adherence.
Stroke survivors adherence rate | 1 month post intervention
  Adherence to the stroke survivors (SS) intervention will be measured by the number of weekly sessions attended (4 total sessions) and total number of hours attended (4 hours) of training completed. Higher number correlates with better outcome.
Change in Post-Study System Usability Questionnaire (PSSUQ) | Baseline, 1 month post intervention
  The Post-Study System Usability Questionnaire will be administered to CPs at the post-treatment evaluation to gather additional data on CARE-CITE usability.
  The PSSUQ is a 19-item survey that measures users' perceived satisfaction with a product or system. Responses are given on a 7-point scale where 1 = strongly agree and 7 = strongly disagree. Responses are averaged to provide a total score between 1 and 7 where low answers indicate greater ease with using the CARE-CITE system.
Carepartner satisfaction | 1 month post intervention
  Carepartner satisfaction will be indicated by scores on a standardized system usability assessment and CARE-CITE module-specific questionnaires. At the end of each of the six modules, carepartners (CP) will be instructed to complete these questions immediately after reviewing a module. Satisfaction will be defined as (1) usefulness of overall content, (2) usefulness of written text, (3) usefulness of videos, (4) ease of use, and (5) acceptability. Each area will be rated using a 5-point Likert type response scale ranging from 1 = strongly disagree to 5 = strongly agree and average scores calculated for each subscale as well as a total score. Total score range 1-5. Higher score correlates with better outcome.

SECONDARY OUTCOMES:
Change in Caregiver Strain assessed by the Caregiver Strain Index (CSI) | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The CSI is a 13-question tool that measures strain related to care provision with binary yes/no answers. There is at least one item for each of the following major domains: Employment, Financial, Physical, Social and Time. Scoring ranges from 0 to 13, with scores of 7 or more indicating greater level of stress.
Change in Bakas Caregiving Outcomes Scale (BCOS) Score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The BCOS is a unidimensional scale based on 10 items and addresses changes in caregiving social functioning, subjective well-being and physical health. Participants respond to statements on a 7-point Likert scale (1=changed for the worst, 7=changed for the best). Total sum of items range from 15-105.
Change in carepartners Family Conflict using Family Caregiver Conflict Scale (FCCS) score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The FCCS is a unidimensional, Likert-type scale composed of 15 items. Each item response is in a Likert-type format with participants indicating their agreement with the item with 1 "not true at all" to 7 "very true." Item scores are summed and higher scores represent higher levels of conflict within a family. Total scores Range 15-105
Change in Family Care Climate Questionnaire - Carepartners (FCCQ-CP) Score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The Family Care Climate Questionnaire (FCCQ) for carepartners is 14-item questionnaire asking about the carepartners' experiences with the strokes survivor in relation to their rehabilitation activities. Each item is rated on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true). Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the carepartner thinks they are providing high autonomy support to the stroke survivor.
Change in Family Care Climate Questionnaire - Stroke Survivor (FCCQ-SS) Score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The Family Care Climate Questionnaire (FCCQ) for stroke survivors is 14-item questionnaire asking about experiences with family members in relation to rehabilitation activities. Each item is rated on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true). Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the stroke survivor perceives receiving high autonomy support from the carepartner.
Change in lower extremity Fugl-Meyer (FM) therapist standardized assessment score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  Total score is sum of 33 items. The possible score range is 0-34. Higher score correlates with less lower extremity (LE) impairment.
Change in stroke survivor gait speed | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The 10-meter walk test will be used, that will look at the time a standardized overground distance. Less time correlates with better outcome.
Change in stroke survivor endurance | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  Will be assessed with the 6-minute walk test, that will look at the distance walked in 6-minutes. It is a measure of aerobic capacity and long-distance walking function. Longer distance correlates with better outcome.
Change in SS Quality of Life using Stroke Impact Scale (SIS) score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  Stroke Impact Scale (SIS) 59-items are broken down into eight domains: strength, hand function, mobility, activities of daily living, emotion, memory, communication, social participation. Domains are scored on a metric of 0 to 100, with higher scores indicating better self-reported health.
Change in Five Times Sit-To-Stand (5TSTS) score | Baseline, 1 week post-intervention, 1 month follow up post-intervention
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Blanton, PT, DPT, Principal Investigator — Emory University
Locations (1):
- Emory Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanton S, Cotsonis G, Brennan K, Song R, Zajac-Cox L, Caston S, Stewart H, Jayaraman A, Reisman D, Clark PC, Kesar T. Evaluation of a carepartner-integrated telehealth gait rehabilitation program for persons with stroke: study protocol for a feasibility study. Pilot Feasibility Stud. 2023 Nov 24;9(1):192. doi: 10.1186/s40814-023-01411-1. PMID 38001523
- [Derived] Blanton S, Cotsonis G, Brenan K, Song R, Zajac-Cox L, Caston S, Stewart H, Jayaraman A, Reisman D, Clark PC, Kesar T. Evaluation of a Carepartner-Integrated Telehealth Gait Rehabilitation Program for Persons with Stroke : Study Protocol for a Feasibility Study. Res Sq [Preprint]. 2023 Apr 14:rs.3.rs-2689016. doi: 10.21203/rs.3.rs-2689016/v1. PMID 37090566